CLINICAL TRIAL: NCT01447251
Title: Assessing the Risk of Developing Type II Diabetes Using Serum Biomarkers in Patients Diagnosed With Obstructive Sleep Apnea
Acronym: OSA & DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWH20110089H
Record Dates: First submitted 2011-09-30; First posted 2011-10-06 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Obstructive Sleep Apnea; Diabetes Mellitus
Keywords: Obstructive Sleep Apnea; Diabetes Mellitus type 2; DM2; OSA; CPAP; continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: Newly Diagnosed/CPAP/NO DM/PreDx DRS (Experimental): patients who have newly-diagnosed obstructive sleep apnea (OSA) requiring continuous positive airway pressure (CPAP) therapy without diabetes and are given the result of the diabetes risk score
  Interventions: Behavioral: PreDx Diabetes Risk Score
- B: Newly Diagnosed/CPAP/NO DM/NO PreDx DRS (Experimental): patients who have newly-diagnosed OSA requiring CPAP therapy without diabetes and are not given the result of the diabetes risk score
  Interventions: Behavioral: PreDx Diabetes Risk Score
- C: Controls (Active Comparator): age, sex, and BMI-matched controls without OSA or diabetes
  Interventions: Behavioral: PreDx Diabetes Risk Score
- D: Controls on CPAP (Active Comparator): age, sex, BMI, and OSA severity matched patients on CPAP therapy for OSA
  Interventions: Behavioral: PreDx Diabetes Risk Score

INTERVENTIONS:
Behavioral: PreDx Diabetes Risk Score — The PreDx DRS measures 7 predictive biomarkers -Adiponectin, C-reactive protein (CRP), Ferritin, Glucose, Insulin, IL-2 and HbA1c, using a proprietary algorithm a risk score in order to calculate a risk score. There are three risk strata, with low risk defined as PreDx DRS <4.5, moderate risk as PreDx DRS ≥4.5 and <8.0, and high risk as PreDx DRS ≥8.0.

SUMMARY:
The investigators plan to recruit 140 patients (35 subjects in each group) over a period of 18 months in a prospective study of matched/paired case-control subjects across the four groups to measure the 5-year risk of developing DM2 in each group and if knowledge of the 5-year risk of developing diabetes will affect continuous positive airway pressure (CPAP) compliance. The study will have four arms: 1) patients who have newly-diagnosed OSA requiring CPAP therapy without diabetes and are given the result of the diabetes risk score; 2) patients who have newly-diagnosed OSA requiring CPAP therapy without diabetes and are not given the result of the diabetes risk score; 3) age, sex, and BMI-matched controls without OSA or diabetes; 4) age, sex, BMI, and OSA severity matched patients on CPAP therapy for OSA. The investigators will document that the patients are compliant with CPAP based on review of SD card data recorded by the CPAP machine. Each patient will have serum drawn for the biomarker panel as well as the standard diagnostic measures of DM2 (oral glucose tolerance test (OGTT) upon enrollment in the study. An Epworth Sleepiness Score, BMI, neck and waist circumference, smoking history, blood pressure, and other standard vital signs will also be collected.

There will be no follow-up of the study subjects in groups 3 and 4 and their participation in this study is completed after Visit 1. Groups 1 and 2 will be followed for 6 months after enrollment to assess whether or not there is any change in CPAP compliance as measured by SD card.

DETAILED DESCRIPTION:
A total of 140 subjects will be recruited (35 subjects with newly-diagnosed obstructive sleep apnea (OSA) without diabetes who will be told their 5-year risk of developing diabetes mellitus type 2 (DM2) prior to starting CPAP therapy, 35 subjects with newly-diagnosed OSA without diabetes who will not be told their 5-year risk of developing DM2 prior to starting continuous positive airway pressure (CPAP) therapy, 35 healthy subjects without OSA or diabetes, and 35 subjects with OSA > 12 months on CPAP therapy). The patients who are newly-diagnosed with OSA will need to be assessed to require CPAP therapy by their treating physician. The investigators will use "A" (ex: A001) before the subject numbers of those subjects newly-diagnosed OSA requiring CPAP therapy without diabetes and are given the result of the diabetes risk score (group 1); and "B" (ex: B001) before the subject numbers of those subjects who have newly-diagnosed OSA requiring CPAP therapy without diabetes and are not given the result of the diabetes risk score (group 2). The investigators will use a "C" (ex: C001) before the subject numbers of the healthy subjects (age, sex, and BMI-matched controls) without OSA or diabetes (group 3). The investigators will use a "D" (ex: D001) before the subject numbers of the (age, sex, BMI, and OSA severity matched) patients on CPAP therapy for OSA (group 4).

Screening Visit:

* Obtain signed Informed Consent document and HIPAA Authorization (research-driven)
* Women of child bearing potential will have a serum pregnancy test (5-10 milliliters (mls), approximately 1-2 teaspoons of blood) (research-driven).
* Review of sleep study data and SD card (flash memory card) data as appropriate to assess for good CPAP compliance as defined by average daily use of >= 4 hours for at least 5 days/week for the 30 days preceding enrollment (standard of care)
* Patients will be told to fast for at least 10 hours prior to Visit 1.

Visit 1 (Day 1):

(see attached Data Collection Form)

* Patients will have the following blood test drawn which include:

  * Biomarker Panel(PreDxTM Diabetes Risk Score),(5-10 mls, approximately 2-4 teaspoons of blood per blood draw)(research-driven) Group 3 & 4 will be shown a sample PreDx Diabetes Risk Report and it will be explained to them. Their report will be mailed to them along with the brochure "A Guide to Understanding Your PreDx Diabetes Risk Score (DRS)".
  * 2-hour OGTT via 2 venipunctures(5-10 mls, approximately 2-4 teaspoons of blood per blood draw)(research-driven)
* Obtain Epworth Sleepiness Score, age, sex, race, height, weight, BMI, neck and waist circumference, smoking history, blood pressure and heart rate (research-driven)
* Patients in group 1 & 2 will be told to fast for at least 10 hours prior to Visit 2.

There will be no follow-up of the study patients in Groups 3 and 4 and their participation in this study is completed after Visit 1.

Visit 1 Follow-Up (Group 1 ONLY)

• Patients will come in and their personalized PreDx Diabetes Risk Report will be explained to them. They will be given the brochure "A Guide to Understanding Your PreDx Diabetes Risk Score (DRS)".

Groups 1 and 2 will have a Visit 2 after 6 months to assess CPAP compliance via SD card review.

Visit 2 (180 days after Visit 1 Follow Up) Groups 1 and 2 only:

(see attached Data Collection Form)

* Patients in Groups 1 and 2 only will be assessed
* Review of sleep study data and SD card (flash memory card) data as appropriate to assess for CPAP compliance over the last 30 days (standard of care)
* Patients will have the following blood test drawn which include:

  o Biomarker Panel (PreDxTM Diabetes Risk Score),(5-10 mls, approximately 2-4 teaspoons of blood per blood draw)(research-driven)
* Obtain Epworth Sleepiness Score, weight, BMI, neck and waist circumference, smoking history, blood pressure and heart rate (research-driven)

Visit 2 Follow-Up (Groups 1 and 2 only):

• Patients will come in and their personalized PreDx Diabetes Risk Report will be explained to them. They will be given the brochure "A Guide to Understanding Your PreDx Diabetes Risk Score (DRS)".

Subjects will be told the results of their 2-hour OGTT by their PCM.

Patients in groups 1 & 2, their participation ends after Visit 2 Follow-Up. Patients in groups 3 & 4, their participation ends after Visit 1.

All patients will receive standard of care treatment regardless of their participation in this research study.

If at any time during the study, the subjects with OSA decided to withdraw from the study, they will be referred to their Primary Care Manager (PCM) to continue standard of care treatment. If the healthy subjects decide to withdraw from the study, no follow up is required. Subjects who are pregnant will be excluded from the study because the changes in a woman's hormones during pregnancy may bias the results of the blood work. Also, women who are breastfeeding may not participate in this study. Study subjects will be told if their Epworth Sleepiness Score is within the normal (0-9) or abnormal (10-24) range; subjects with abnormal Epworth scores will be instructed to follow-up with their PCM. If the healthy subjects decide to withdraw from the study, no follow up is required. If a subject is diagnosed as being diabetic or pre-diabetic as part of this study, they will be referred to their PCM for standard of care treatment. If patients are withdrawn from the study, no further testing as part of this study is required. If patients decide to withdraw from the study, any remaining portion of their blood sample will be destroyed. However, any data already obtained by researchers from their sample will continue to be used for research purposes discussed in this protocol.

Diabetes Risk Score (Pre Dx DRS) The PreDx DRS test sample will be collected as follows: Tethys Biosciences will send prepared collection kits and packing materials. Blood will be drawn in 2 tubes containing 8.5 mL and 4 mL respectively by lab personnel after the patient has been fasting for 10 hours, requiring one venipuncture. The collection kit will be assigned a de-identified number. We will keep a locked master list of the code number associated with the patient's identification. The collected blood will be processed and stored according to manufacturers'specifications. The lab kits will be shipped to Tethys Biosciences within 7 days. From the sample, Tethys Bioscience will measure 7 predictive biomarkers -Adiponectin, C-reactive protein (CRP), Ferritin, Glucose, Insulin, IL-2 and HbA1c. Using a proprietary algorithm a risk score is calculated. In order to calculate the risk score, Tethys will need the patients' dates of birth and gender in addition to the fasting blood sample. The PreDx DRS model provides a continuous measure of risk of progressing to DM2 within five years. There are three risk strata, with low risk defined as PreDx DRS <4.5, moderate risk as PreDx DRS ≥4.5 and <8.0, and high risk as PreDx DRS ≥8.0. Tethys Bioscience will send the results of the PreDx DRS test to the Clinical Research Coordinator.

The Tethys Biosciences Clinical Laboratory is Clinical Laboratory Improvement Amendments (CLIA) certified and will use these procedures when processing Laboratory specimens mentioned in this research project.

This test was developed and its performance characteristics determined by the Tethys Clinical Laboratory. The results are not intended to be used as the sole means for clinical diagnosis or patient management decisions.

ELIGIBILITY:
Inclusion:

* Tricare beneficiaries (military insurance) eligible for care at Nellis AFB.
* Male or Female > 18 years old
* Groups 1 and 2: newly diagnosed with OSA and determined to need continuous positive airway pressure (CPAP) therapy by their treating physician
* Group 4: known diagnosis of obstructive sleep apnea (OSA) treated with CPAP therapy for 12-24 months with demonstrated compliance after review of SD card
* Tricare Beneficiaries

Exclusion:

* Diagnosed as being diabetic by having a positive oral glucose tolerance test for diabetes
* Pregnant or breastfeeding
* Groups 1 and 2: being diagnosed for OSA for greater than one month
* Groups 1, 2, and 4: being diagnosed for OSA but not needing CPAP therapy
* Groups 1, 2, and 4: treatment of OSA with CPAP therapy but CPAP machine does not have SD card
* Group 3: being diagnosed with OSA
* Group 4: being diagnosed for OSA for less than one year
* All non-English speaking subjects or those who do not demonstrate the ability to understand the study or the willingness to sign the written informed consent document will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with a change in their seven serum biomarker panel results | 12 months

SECONDARY OUTCOMES:
Number of participants with increased Continuous Positive Airway Pressure (CPAP)Compliance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Walpole, D.O, Capt, Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis AFB
Locations (1):
- Mike O'Callaghan Federal Hospital/Nellis AFB, Las Vegas, Nevada, United States